CLINICAL TRIAL: NCT00435799
Title: Treatment of Keratectasia With Collagen Cross-Linking (CCL) at the Eye Departments of the University Hospital, North Norway in Tromsø and Ullevål University Hospital in Oslo
Brief Title: Evaluating Collagen Cross-Linking (CCL) Treatment in Norway
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: ALEKSANDAR STOJANOVIC, MD, University Hospital of North Norway
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNN-UUS-CCL07
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2007-01

CONDITIONS: Keratoconus
Keywords: keratoconus; corneal cross-linking; riboflavine; ultraviolet type A rays (UVA)
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking; Riboflavin

ARMS (1):
- A (Active Comparator)
  Interventions: Procedure: corneal cross-linking (CCL); Drug: Riboflavin/dextran eyedrops; Device: UV-X system

INTERVENTIONS:
Procedure: corneal cross-linking (CCL)
  Other Names: Riboflavine; UVX
Drug: Riboflavin/dextran eyedrops
Device: UV-X system

SUMMARY:
The purpose of this study is to assess safety, efficacy and stability of riboflavin-UV induced cross-linking of corneal collagen in reducing the progression of keratecatasia and in improving visual acuity. This is the first Norwegian study concerning CCL.

DETAILED DESCRIPTION:
The technique of corneal collagen cross-linking consists of photopolymerization of stromal fibers by combined action of a photosensitizing substance, riboflavin and ultraviolet type A rays (UVA) from a solid-state UVA Source. Photopolymerization increases the rigidity of corneal collagen and its resistance to keratectasia. It has been used to stop progression of keratectasia.

Corneal transplantation has been the only available option so far for treatment for keratectasia in its advanced stage in Norway. The method of CCL using riboflavin and UV light is technically simple and much less invasive than corneal transplantation and it treats and prevents the underlying pathophysiological mechanism. It also does not reduce the chances for a successful corneal transplantation, in case that would still be necessary after CCL.

The purpose of this study is to assess safety, efficacy and stability of riboflavin-UV induced cross-linking of corneal collagen in reducing the progression of keratecatasia and in improving visual acuity. This is the first Norwegian study concerning CCL.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 45 years
2. Progressive keratectasia (primary or secondary) in an advanced stage
3. Decreased best corrected visual acuity bellow 20/40, which cannot be further improved by use of soft contact lenses
4. Rigid contact lenses are either not tolerated or do not improve visual acuity
5. No previous eye surgery (except for laser refractive surgery)
6. All patients must provide written informed consent to become a study subject
7. Subjects able to return for scheduled follow-up examinations according to this protocol

Exclusion Criteria:

1. Corneal thickness < 400 µm at thinnest position
2. Keratometric - readings above 60 diopters
3. Other active ocular disease than keratectasia
4. Herpes keratitis
5. Previous ocular surgery (other than laser refractive surgery)
6. Patients who were immunocompromised, pregnant or who had atopic syndrome, connective tissue or autoimmune disease
7. Patients with known sensitivity to study medication
8. Subjects with intraocular pressure > 23 mmHg by Goldmann applanation tonometry, a history of glaucoma, or glaucoma suspects
9. Subjects who intent to participate in other ophthalmic clinical trails during this clinical investigation

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
1 Efficacy will be evaluated based on: a. reduction of keratometry (curvature) values, b. improvement in distance best spectacle corrected visual acuity (BSCVA) and c. improvement in patients visual disturbances.
2 Stability of the treatment will be evaluated based on keratometry and on manifest refraction spherical equivalent (MRSE).
3 Safety will be evaluated based on the changes in distance best spectacle corrected visual acuity (BSCVA).

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Stojanovic, MD, Principal Investigator — Eye dpt, University Hospital of North Norway
Locations (2):
- Norway (2):
  - Eye dpt, Ullevål University Hospital, Oslo, Oslo County
  - Eye dpt, University Hospital North Norway, Tromsø, Tromsø